CLINICAL TRIAL: NCT07088289
Title: Virtual Reality Mindfulness Intervention for Supporting People With HIV and Substance Use
Brief Title: VR Mindfulness for People With HIV and Substance Use
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Responsible Party: Principal Investigator, Audrey Hai, Assistant Professor, Tulane University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-949; R21DA061682 (NIH)
Record Dates: First submitted 2025-07-19; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: HIV; Substance Use (Drugs, Alcohol)
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VR mindfulness (Experimental): Participants in this arm will receive a virtual reality (VR) mindfulness intervention named TRIPP. TRIPP is a commercially available VR mindfulness app designed to promote relaxation, focus, and emotional well-being through immersive, guided experiences. The app combines visual and auditory stimulation, breathwork, meditation, and interactive elements to help users reduce stress and improve mood.
  Interventions: Behavioral: TRIPP

INTERVENTIONS:
Behavioral: TRIPP — In this study, participants will use TRIPP with a VR headset at home, engaging in short mindfulness sessions 3+ times per week for 4-12 weeks.

SUMMARY:
The goal of this clinical trial is to explore whether a virtual reality (VR) mindfulness app is acceptable, appropriate, and feasible for supporting people with HIV and substance use problems.

Participants will:

* Use a VR headset with a mindfulness app at home;
* Complete three online surveys over three months;
* Take part in an individual interview or focus group to share their experiences.

ELIGIBILITY:
Inclusion Criteria:

* Able to speak, read, and write in English
* Aged 18 years or older
* Diagnosed with HIV
* Currently prescribed ART therapy
* Reporting moderate to high risk related to alcohol, opioids, nicotine, cannabis, or stimulant use (score of 4 or higher on the Alcohol, Smoking, and Substance Involvement Screening Test - ASSIST). Participants may also use other substances, but the primary risk must fall within these categories, as these have the strongest research support for mindfulness-based interventions.
* Having stable housing that allow using VR safely
* Willing to provide contact information for at least one person whom the study team can reach if the participant becomes unreachable after repeated attempts

Exclusion Criteria:

* Living in institutionalized settings or unsheltered
* Terminal illness with a life expectancy of less than 6 months
* Planning to move out of the area in the next eight weeks
* Engaging in regular mindfulness practice outside of TRIPP
* Experiencing fear of closed spaces or unable to tolerate wearing a VR headset (verified during orientation session)
* Having visual or auditory impairments or severe physical disabilities that hinder VR use, history of seizures, severe cognitive impairment, severe motion sickness, severe unmanaged psychiatric symptoms, or currently pregnant
* Participants without home internet access will not be excluded and will be provided either funding for internet service or VR headsets preloaded with TRIPP sessions for offline use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Intervention acceptability as measured by the Acceptability of Intervention Measure | One-month follow-up
  The Acceptability of Intervention Measure is a 4-item scale that assesses the extent to which participants find the intervention agreeable or satisfactory. Items are rated on a 5-point Likert scale ranging from 1 (Completely disagree) to 5 (Completely agree). Scores are averaged to create a total score, with higher scores indicating greater perceived acceptability of the intervention. Example items include: "I like [intervention]" and "[intervention] meets my approval."
Intervention appropriateness as measured by the Intervention Appropriateness Measure | One-month follow up
  The Intervention Appropriateness Measure is a 4-item scale designed to assess how suitable or relevant the intervention is for the target population. Each item is rated from 1 (Completely disagree) to 5 (Completely agree), and a total score is calculated by averaging responses. Higher scores reflect a stronger belief that the intervention is appropriate for the individual's needs or situation. Example items include: "[intervention] seems like a good match" and "[intervention] seems suitable."
Intervention feasibility as measured by the Feasibility of Intervention Measure | One-month follow up
  The Feasibility of Intervention Measure includes 4 items that measure how practical and doable the intervention seems from the participant's perspective. Participants respond on a 5-point scale from 1 (Completely disagree) to 5 (Completely agree), with higher average scores indicating greater perceived feasibility. Example items include: "[intervention] seems implementable" and "[intervention] seems easy to use."

SECONDARY OUTCOMES:
Intervention engagement as measured by VR mindfulness app use frequency | From enrollment to the end at 12 weeks.
  Engagement with the intervention will be measured by the frequency of VR mindfulness app use, as recorded by the TRIPP app. The system captures the number of times participants launch and complete mindfulness sessions during the study period. Higher session counts reflect greater engagement with the intervention. There is no maximum score, and a higher number of sessions indicates more frequent use of the app.

IPD SHARING:
Plan to Share IPD: Yes